CLINICAL TRIAL: NCT01889550
Title: Use of eHealth in Communication With Patients About Prenatal Diagnosis. An Intervention Study Carried Out in a Highly Specialised Unit for Obstetrics
Brief Title: Use of eHealth in Communication With Patients About Prenatal Diagnosis
Acronym: HIIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mette Maria Skjoeth, PhD Student, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HIIP
Record Dates: First submitted 2013-06-19; First posted 2013-06-28 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Downs Syndrome; Health Knowledge, Attitudes, Practice
Keywords: Screening; Downs syndrome; Informed choice; eHealth
MeSH Terms: conditions — Down Syndrome; Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Access to the website www.graviditetsportalen.dk (Active Comparator): The website www.graviditetsportalen.dk contains information about the screeningtest for Downs syndrome. The website uses both text, video and animated graphics.
  Interventions: Behavioral: Access to the website www.graviditetsportalen.dk
- Access to the website www.ouh.dk (Placebo Comparator): Access to the usual information from the hospital website
  Interventions: Behavioral: Access to the website www.ouh.dk

INTERVENTIONS:
Behavioral: Access to the website www.graviditetsportalen.dk — The website www.graviditetsportalen.dk contains information about the screeningtest for Downs syndrome. The website uses both text, video and animated graphics.
  Other Names: Website
  Arms: Access to the website www.graviditetsportalen.dk
Behavioral: Access to the website www.ouh.dk — Access to the usual information from the hospital website
  Arms: Access to the website www.ouh.dk

SUMMARY:
The research aims at generating new knowledge about ways to inform pregnant women about prenatal screening for Downs syndrome.

The overall purpose of this project is to increase pregnant women's knowledge of prenatal screening for Downs syndrome, and thereby an option to make an informed choice. The project is planned as a research into whether the use of an eHealth solution (in this project an interactive website) may be an appropriate intervention for pregnant women.

DETAILED DESCRIPTION:
Prenatal screening and diagnosis is testing for diseases or rare conditions in the fetus before birth. The aim is to assist the pregnant women to make their own decisions, and neutral and adequate counseling is a prerequisite during prenatal diagnosis. To make an informed choice, the pregnant women must be informed about the benefits and potential disadvantages of prenatal diagnosis and with this background be able to make a comprehensive evaluation, where ethical values will have a high impact.

The overall purpose of this project is to increase pregnant women's knowledge of prenatal screening for Downs syndrome, and thereby an option to make an informed choice. The project is planned as a research into whether the use of an eHealth solution (in this project an interactive website) may be an appropriate intervention for pregnant women.

Methods:

Part one consists of an identification of the problem

Part two consists of developing a website with relevant information about prenatal screening for Downs syndrome.

Part three is an effect measurement. The effect of the intervention is measured through a randomized controlled trail in which the essentials of the measurement will be the pregnant women's knowledge and behavior in relation to prenatal diagnosis. Twice 300 pregnant women will be included in the project.

Results:

The research aims at generating new knowledge about ways to inform pregnant women about prenatal diagnosis and prenatal screening. The expected results are:

* Higher knowledge about prenatal diagnosis for the pregnant women.
* Less difficulty in making an informed choice for the coming parents.
* Easy access to high quality information.
* Equity in access to high quality information.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women participating in screening for Downs syndorme

Exclusion Criteria:

* Respondents who do not speak, read and understand Danish.
* Respondents who have opted out of health care services and prenatal diagnosis.
* Reespondenter who do not wish to participate.
* Respondents under 18 years.
* Respondents with a strong suspicion of threatening abortion
* Respondents whom are vulnerable
* Respondents with a late referral

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1150 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Multidimensional measure of informed choice (MMIC) | Participants will be asked to compleete the questionnaire in an expected average of 6 weeks after having had the nuchal translucency scan.
  Questionnaire for assessing knowledge of prenatal screening for Downs syndrome

SECONDARY OUTCOMES:
Decisional Conflict Scale | Participants will be asked to compleete the questionnaire in an expected average of 6 weeks after having had the nuchal translucency scan.
WHO well-being index | Participants will be asked to compleete the questionnaire in an expected average of 6 weeks after having had the nuchal translucency scan.
Cambridge Worry Scale | Participants will be asked to compleete the questionnaire in an expected average of 6 weeks after having had the nuchal translucency scan.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Maria Skjoeth, PhD Student, Principal Investigator — Odense University Hospital, Department of Gynaecology and Obstetrics, University of Southern Denmark, Institute of Clinical research, Research Unit of Gynaecology and Obstetrics; Jan Stener Joergensen, Associate professor, Study Chair — Odense University Hospital, Department of Gynaecology and Obstetrics, University of Southern Denmark, Institute of Clinical research, Research Unit of Gynaecology and Obstetrics; Claus Duedal Pedersen, Head of Innovation Unit, Study Chair — Odense University Hospital, The LEAN and Innovation Unit; Eva Draborg, Associate professor, Study Chair — University of Southern Denmark, Centre of Health Economics Research - Institute of Public Health; Helle Ploug Hansen, Professor, Study Chair — University of Southern Denmark, The Institute of Public Health
Locations (1):
- Odense University Hospital, Department of Gynaecology and Obstetrics, Odense, Region Syddanmark, Denmark